CLINICAL TRIAL: NCT04979403
Title: Efficacy of a Psychologically-Informed Physiotherapy Intervention in Patients With Chronic Low Back Pain With a High Level of Psychosocial Factors: a Feasibility and Pilot Randomized Clinical Trial
Brief Title: Efficacy of Two Physiotherapy's Approaches in Chronic Low Back Pain: Is Addressing Psychosocial Factors Beneficial?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale (Other); Fonds de la Recherche en Santé du Québec (Other Government); Ordre professionnel de la physiothérapie du Québec (Unknown)
Responsible Party: Principal Investigator, Hugo Massé-Alarie, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-2227
Record Dates: First submitted 2021-06-14; First posted 2021-07-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain, Recurrent
Keywords: Chronic low back pain; Psychosocial factors; Physiotherapy; Interventions
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: It is a feasibility and pilot randomized clinical trial. Participants will be assigned to either the psychologically-informed physiotherapy intervention or to the usual care in physiotherapy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care in physiotherapy (Active Comparator): The usual care group will receive interventions recommended by clinical guidelines: education on the nature of LBP, advice to stay active and to continue usual activities, specific exercise programs combined with orthopedic manual therapy.
  Interventions: Other: Physiotherapy
- Psychologically-informed physiotherapy intervention (Experimental): The psychologically-informed physiotherapy group will receive the control intervention enhanced with specific interventions targeting psychosocial factors (e.g., positive reinforcement, mindfulness-based stress reduction, diaphragmatic breathing, graded exposure). Most of these techniques are efficient to mitigate the impact of psychological factors such as anxiety and fear of movement. To standardize the psychologically-informed physiotherapy approach, physiotherapists will receive a two-day training course by a physiotherapist expert with this approach in chronic pain conditions (Alain Gaumond).
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Participants from each group will receive 8 intervention sessions (45 min) over 11 weeks by a physiotherapist. For both groups, each intervention will be tailored to the patient's profile and the choice of interventions and parameters will be at the judgment of the physiotherapist.

SUMMARY:
Low back pain is presently the first cause of disability worldwide. The most recommended interventions by clinical guidelines are exercises and cognitive behavioral therapy although the effect is modest. However, no approach is superior when given to a heterogeneous group of subjects with chronic low back pain (CLBP). This is probably due to the multiple factors associated with CLBP which are biophysical, psychological and social. Thus, each patient presents with a unique profile of factors contributing to their pain and could benefit from an approach tailored to their profile. In other words, it is crucial to identify the right treatment, for the right person, at the right moment. For example, the presence of important psychological factors such as anxiety and depression are risk factors for low back pain to develop and persist over time. The main aim of this project is to determine the feasibility to perform a large clinical trial comparing the efficacy of a two physiotherapy's approaches to treat CLBP (i.e., a psychologically-informed physiotherapy intervention compared to usual physiotherapy) in patients with CLBP presenting a high level of psychological factors.

DETAILED DESCRIPTION:
Low back pain is presently the first cause of disability worldwide. The most recommended interventions by clinical guidelines are exercises and cognitive behavioral therapy although the effect is modest. However, no approach is superior when given to a heterogeneous group of subjects with chronic low back pain (CLBP). This is probably due to the multiple factors associated with CLBP which are biophysical, psychological and social. Thus, each patient presents with a unique profile of factors contributing to their pain and could benefit from an approach tailored to their profile. In other words, it is crucial to identify the right treatment, for the right person, at the right moment. For example, the presence of important psychological factors such as anxiety and depression are risk factors for low back pain to develop and persist over time. Empowerment of physiotherapists and patients on the optimal management of psychosocial factors, in addition of the usual care delivered in physiotherapy, may be a potent strategy to improve the treatment effect especially with patients presenting a complex clinical profile. This empowerment may be done through psychologically-informed physiotherapy, an approach incorporating strategies from cognitive behavioral therapy into the physiotherapy usual practice. However, the feasibility to perform a clinical trial including psychologically-informed physiotherapy in the context of the Quebec's healthcare system remains to be verified.

The main aim of this project is to determine the feasibility to perform a pilot randomised controlled trial testing the efficacy of a psychologically-informed physiotherapy intervention in CLBP patients with a high level of psychosocial factors compared to usual physiotherapy. Specific aims are related to feasibility (1) and sample size estimation (2):

1. To test (a) strategies to recruit participants with high level of psychosocial factors and physiotherapists (PT) (recruitment rate and retention), (b) the physiotherapists and participants adherence to intervention, (c) the risk of contamination between treatment sites and (d) specific challenges;
2. To gather data to estimate the required sample size for a future full-scale randomized clinical trial using physical functioning as main outcome, and pain intensity, quality of life, fear of movement, catastrophizing, self-efficacy, pain pressure threshold, exercise-induced hypoalgesia and temporal summation as additional outcomes.

The hypothesis is that this project will be feasible in terms of recruitment for both patients (~30) and PT (6-8), will show good patients and physiotherapists' adherence to intervention and low contamination between treatment sites. An improvement for all pain-related outcomes in both groups, but more in the psychologically-informed physiotherapy group, is also expected.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic low back pain (> 3 months)
* High level of psychosocial factors (a high level using the Start Back Screening Tool, i.e., cut-off of at least 4 points (total score) and at least 4 points (sub-score with questions 5 to 9)).

Exclusion Criteria:

* Non-musculoskeletal conditions causing low back pain (e.g., neoplasia, infection)
* Neuropathic conditions (e.g., radiculopathy).
* Currently in litigation with paying agencies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of participants | Baseline
  The number of participants contacted divided by the number of participants recruited.
Physiotherapists adherence to intervention | Week 6
  Physiotherapists will complete a list of interventions used after each interventions (8 interventions on period of 6 weeks).
Risk of contamination between treatment sites | Week 6
  The list of interventions used by physiotherapists at each site will be compared to evaluate the risk of contamination between treatment sites.
Specific challenges | Through data collection completion, an average of 1 year
  Using semi-structured interview with the physio.
Retention of participants | Baseline, when a participant drop out
  The number of participants who completed the study divided by the number of participants that were recruited.
Participants adherence to intervention | Week 6
  Participants will measure their adherence to intervention on a Numeric Rating Scale from 0 (not adherent at all) to 10 (completely adherent).

SECONDARY OUTCOMES:
Physical functioning (ODI) | Baseline, Weeks 6, 12 and 24
  The Oswestry Disability Index (ODI) is a self-completed questionnaire on estimated disability including 10 questions rated on a 6-item scale, from 0 (no disability) to 5 points (maximal disability).
Pain intensity (NRS) | Baseline, Weeks 6, 12 and 24
  The Numeric Rating Scale (NRS) is an 11-point scale used to score the intensity of pain in the last week ranging from 0 (no pain) to 10 (worst imaginable pain).
Quality of life (SF-12) | Baseline, Weeks 6, 12 and 24
  The 12-Item Short Form Survey is a self-completed questionnaire counting 12 questions on eight mental and physical health domains. The score is calculated by a specific calculator that compares the score to the general population.
Fear of movement (TSK-11) | Baseline, Weeks 6, 12 and 24
  The Tampa Scale of Kinesiophobia is a self-completed questionnaire used to assess fear of movement using 11 questions on a 4-point scale ranging from 1 (strongly disagree, low level of kinesiophobia) to 4 (strongly agree, high level of kinesiophobia).
Catastrophizing thoughts (PCS) | Baseline, Weeks 6, 12 and 24
  The Pain Catastrophizing Scale (PCS) is a self-completed questionnaire of 13 questions measuring catastrophizing thoughts contributing to pain on a 5-point scale ranging from 0 (not at all, low level of catastrophizing thoughts) to 5 (all the time, high level of catastrophizing thoughts).
Self-efficacy (CPSES) | Baseline, Weeks 6, 12 and 24
  The Chronic Pain Self-Efficacy Scale (CPSES) (short form) is a self-completed questionnaire of 6 questions measuring self-efficacy on a 10-point scale from 0 (not at all confident, low self-efficacy) to 10 (completely confident, high self-efficacy).
Participant's expectations | Baseline, Weeks 6, 12 and 24
  Participant's expectations regarding treatment will be measured with a self-completed questionnaire of three 7-level Likert questions on pain, physical functioning and participation ranging from 0 (way better) to 6 (way worst).
Central Sensitization (CSI) | Baseline, Weeks 6, 12 and 24
  The Central Sensitization Index (CSI) is a self-completed questionnaire of 9 questions measuring central sensitization on a 5-point scale from 0 (never, low level of central sensitization) to 5 (always, high level of central sensitization).
Global rating of change (GRC) | Baseline, Weeks 6, 12 and 24
  The Global rating of change (GRC) is a 11-point scale ranging from -5 (a great deal worst) to 5 (a great deal better) to measure the perceived change oh health status after the intervention.
Pain pressure threshold | Baseline, Week 6
  Pain pressure thresholds will be measured at 3 sites (L4-L5 paravertebral, upper and lower legs) using a digital algometer before and after an exercise of wrist flexion (maintaining 25% of the maximal voluntary contraction activity during 4 minutes) to test the exercise-induced hypoalgesia paradigm.
Temporal summation | Baseline, Week 6
  Temporal summations will be measured at 3 sites (L4-L5 paravertebral, upper and lower legs) using a pinprick before the exercise of wrist flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Massé-Alarie, PhD, Principal Investigator — Laval University
Locations (1):
- Cirris (Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (of all primary and secondary outcomes) will be available in a supplementary table when publishing the results of the study.
Supporting Information: Study Protocol
Time Frame: The data will become available when the results of the study will be published (around winter 2023) for an unlimited period.
Access Criteria: The data will become available when the results of the study will be published (around winter 2023) for an unlimited period.

REFERENCES:
- [Result] Masse-Alarie H, Desgagnes A, Cote-Picard C, Liberty O, Langevin P, Piche M, Tousignant-Laflamme Y. Comparisons of the effects of psychologically-informed and usual physiotherapy on pain sensitivity in chronic low back pain: an exploratory randomized controlled trial. Arch Physiother. 2025 Feb 17;15:32-41. doi: 10.33393/aop.2025.3323. eCollection 2025 Jan-Dec. PMID 39974748
- [Result] Desgagnes A, Cote-Picard C, Gaumond A, Langevin P, Piche M, Page G, Pinard AM, Tousignant-Laflamme Y, Masse-Alarie H. Efficacy of a Psychologically-Informed Physiotherapy Intervention in Patients with Chronic Low Back Pain at High Risk of Poor Prognosis: A Pilot and Feasibility Randomized Controlled Trial. Physiother Can. 2024 May 8;76(2):163-174. doi: 10.3138/ptc-2023-0038. eCollection 2024 May. PMID 38725600